CLINICAL TRIAL: NCT00693186
Title: An Open-label, Randomised, Controlled, Multi-centre Study of the Immunogenicity and Safety of a Booster Dose of Two Different Hepatitis B Vaccines to Explore the Anamnestic Immune Response in Healthy 4 to 7 Year-old Children Previously Vaccinated at About 3, 5 and 11 to 13 Months of Age With Either HEXAVAC® or INFANRIX®-HEXA
Brief Title: A Study to Assess the Anamnestic Immune Response in Healthy 4 to 7 Year-old Children After a Primary Vaccination Series With Either HEXAVAC® or INFANRIX®-HEXA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HXV01C
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — Hepatitis B Vaccines; Engerix-B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Biological: HBVaxPRO® 5 µg / 0.5 mL
- 2 (Experimental)
  Interventions: Biological: Engerix B® 10 µg / 0.5 mL

INTERVENTIONS:
Biological: HBVaxPRO® 5 µg / 0.5 mL — 5 µg / 0.5 mL
  Arms: 1
Biological: Engerix B® 10 µg / 0.5 mL — 10 µg
  Arms: 2

SUMMARY:
Primary objective:

* To describe in subjects vaccinated with 3 doses of HEXAVAC® or 3 doses of INFANRIX®-HEXA during the first two years of life the percentage of subjects with an anti-HBs antibody titre ≥10 mIU/mL 1 month after a booster dose of either HBVaxPRO® 5 µg or Engerix B® 10 µg .

Secondary objectives:

* Additional immunogenicity assessments
* Standard safety assessment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy child of 4 to 7 years of age of either gender,
* Child vaccinated with 2 doses of HEXAVAC® during the first 6 months of life and with a 3rd dose of HEXAVAC® before the end of the second year of life or Child vaccinated with 2 doses of INFANRIX®-HEXA during the first 6 months of life and with a 3rd dose of INFANRIX®-HEXA before the end of the second year of life,
* Informed consent form signed by the parent(s) or by the legal representative.
* Parent(s) or legal representative able to understand and comply with the study procedures.

Exclusion Criteria:

* Any recent (<=3 days) history of febrile illness prior to vaccination,
* Receipt of more than 3 doses of any Hepatitis B containing vaccine, either alone or in any combination,
* History of clinical or serological-confirmed diagnosis of infection due to hepatitis B,
* History or current close contact with known carriers of hepatitis B virus,
* Prior known sensitivity/allergy to any component of the study vaccines,
* Any known blood dyscrasias, leukemia, lymphomas of any type, or other malignant neoplasms affecting the haematopoietic and lymphatic systems,
* Any severe thrombocytopenia or any other coagulation disorder that would contraindicate intramuscular injection,
* Any immune impairment or humoral/cellular deficiency or depressed immunity,
* Any recent (<=30 days) long-term (>=14 days) administration of systemic corticosteroids given daily or on alternate days at >=20 mg/day prednisone equivalent or scheduled administration through Visit 2,
* Any receipt (<=3 months) of immunoglobulins or blood-derived products, or scheduled administration through Visit 2,
* Any recent (<=14 days) receipt of an inactivated vaccine or scheduled administration through Visit 2,
* Any recent (<=28 days) receipt of a live vaccine or scheduled administration through Visit 2

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 410 (Actual)
Dates: Start 2008-10 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with anti-HBs antibody titres >=10 mIU/mL measured at 1 month post-booster dose | 28 to 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (5):
- Italy (5):
  - Unità Operativa Semplice di Epidemiologia (UOSE), Quarto, Napoli
  - Azienda per i Servizi Sanitari n. 5 "Bassa Friulana", Latisana, Udine
  - Ospedale Maggiore di Modica - Via Resistenza Partigiana (c/o Ospedale Maggiore), Modica
  - AUSL n. 7 di Ragusa Servizio di Epidemiologia Via G. Di Vittorio 59/c, Ragusa
  - Dipartimento di Prevenzione Servizio di Igiene Pubblica, Sassari

REFERENCES:
- [Derived] Zanetti A, Parlato A, Romano L, Desole MG, Ferrera G, Giurdanella F, Zuliani M, Richard P, Thomas S, Fiquet A. Challenge with a hepatitis B vaccine in two cohorts of 4-7-year-old children primed with hexavalent vaccines: an open-label, randomised trial in Italy. Vaccine. 2012 Aug 24;30(39):5770-5. doi: 10.1016/j.vaccine.2012.06.078. Epub 2012 Jul 9. PMID 22789511